CLINICAL TRIAL: NCT00637637
Title: Radiation Therapy in Combination With Indinavir / Ritonavir (Crixivan / Norvir) for the Treatment of Brain Metastases: a Randomized Phase II Study
Brief Title: External-Beam Radiation Therapy With or Without Indinavir and Ritonavir in Treating Patients With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncology Institute of Southern Switzerland (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: IOSI-RO0402; CDR0000587517 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-03-14; First posted 2008-03-18 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-12

CONDITIONS: Cancer
Keywords: tumors metastatic to brain; stage IV adenoid cystic carcinoma of the oral cavity; stage IV adrenocortical carcinoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV anal cancer; stage IV basal cell carcinoma of the lip; stage IV bladder cancer; stage IV borderline ovarian surface epithelial-stromal tumor; stage IV breast cancer; stage IV childhood anaplastic large cell lymphoma; stage IV childhood Hodgkin lymphoma; stage IV childhood large cell lymphoma; stage IV childhood liver cancer; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV chronic lymphocytic leukemia; stage IV colon cancer; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV esophageal cancer; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV follicular thyroid cancer; stage IV gastric cancer; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV hypopharyngeal cancer; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV laryngeal cancer; stage IV lip and oral cavity cancer; stage IV lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the oropharynx; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV mycosis fungoides/Sezary syndrome; stage IV nasopharyngeal cancer; stage IV non-small cell lung cancer; stage IV oropharyngeal cancer; stage IV ovarian epithelial cancer; stage IV pancreatic cancer; stage IV papillary thyroid cancer; stage IV paranasal sinus and nasal cavity cancer; stage IV penile cancer; stage IV prostate cancer; stage IV rectal cancer; stage IV renal cell cancer; stage IV salivary gland cancer; stage IV small lymphocytic lymphoma; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV endometrial carcinoma; stage IV verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the oral cavity; stage IVB vulvar cancer; stage IV Wilms tumor; stage IVB cervical cancer; stage IVB vaginal cancer; metastatic adult malignant fibrous histiocytoma of bone; metastatic childhood malignant fibrous histiocytoma of bone; metastatic gastrointestinal carcinoid tumor; metastatic parathyroid cancer; metastatic pheochromocytoma; metastatic squamous neck cancer with occult primary squamous cell carcinoma; metastatic squamous neck cancer with occult primary; metastatic transitional cell cancer of the renal pelvis and ureter; disseminated neuroblastoma; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; tongue cancer
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Adrenocortical Carcinoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Anus Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Lymphocytic, Chronic, B-Cell; Colonic Neoplasms; Lymphoma, T-Cell, Cutaneous; Esophageal Neoplasms; Esthesioneuroblastoma, Olfactory; Adenocarcinoma, Follicular; Stomach Neoplasms; Lymphoma, Follicular; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Mycosis Fungoides; Sezary Syndrome; Nasopharyngeal Neoplasms; Carcinoma, Non-Small-Cell Lung; Oropharyngeal Neoplasms; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Thyroid Cancer, Papillary; Penile Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Endometrial Neoplasms; Vulvar Neoplasms; Wilms Tumor; Uterine Cervical Neoplasms; Vaginal Neoplasms; Histiocytoma, Malignant Fibrous; Parathyroid Neoplasms; Pheochromocytoma; Tongue Neoplasms | interventions — Indinavir; Ritonavir; Radiotherapy

INTERVENTIONS:
Drug: indinavir sulfate
Drug: ritonavir
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Indinavir and ritonavir may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether external-beam radiation therapy is more effective with or without indinavir and ritonavir in treating patients with brain metastases.

PURPOSE: This randomized phase II trial is studying external-beam radiation therapy alone to see how well it works compared to external-beam radiation therapy given together with indinavir and ritonavir in treating patients with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy, in terms of time to treatment failure at CNS level and 4-months treatment failure rate, in patients with brain metastases treated with external-beam radiotherapy in combination with indinavir sulfate and ritonavir versus external-beam radiotherapy alone.
* Prospectively investigate the efficacy of a potentially antiangiogenic agent, indinavir sulfate.
* Investigate the antineoplastic activity of indinavir sulfate in combination with ionizing radiation in cancer patients with metastatic disease to the brain.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy to the brain once daily, 5 days a week for 2 weeks (10 doses total). Patients also receive oral indinavir sulfate and oral ritonavir twice daily for 35 days beginning at day 1 of radiotherapy.
* Arm II: Patients undergo radiotherapy to the brain once daily, 5 days a week for 2 weeks (10 doses total).

Patients complete quality of life questionnaires, including QOL-30 and the Mini Mental Status Examination, at baseline, 2 weeks after completion of radiotherapy, and at 1 and 3 months after completion of study treatment.

After completion of study treatment, patients are followed periodically for at least 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic cancer with brain metastases

  * Biopsy of brain metastases is not required
* All cancer types allowed, except for the following:

  * Prostatic adenocarcinoma
  * Sarcoma
  * Melanoma
  * Germ cell carcinoma,
  * Small-cell lung cancer
* Measurable disease by MRI of the brain
* Not requiring immediate surgical decompression (may qualify after surgery, if remaining measurable brain lesions)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2 (corresponds to recursive partitioning analysis groups I or II)
* Life expectancy > 4 months
* Able to understand the aim of trial and to comply with follow-up
* No HIV seropositivity

PRIOR CONCURRENT THERAPY:

* Prior dexamethasone allowed provided it is tapered before initiation of study radiotherapy
* Not requiring cytotoxic treatment within 3 months after study radiotherapy
* At least 1 week since prior and no concurrent phenytoin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure in the brain (TTF) as determined by the radiological response rate
Overall survival (OS)
Radiological volumetric response to treatment
Local intracranial disease progression at 4 months
Progression-free survival at 6 months

SECONDARY OUTCOMES:
Improvement of symptoms
Time to symptom relapse or symptom progression
Duration of use of steroids
Duration of use of anticonvulsive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Ilja Ciernik, MD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (3):
- Switzerland (3):
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Oncology Institute of Southern Switzerland - Lugano, Lugano
  - UniversitaetsSpital Zuerich, Zurich